CLINICAL TRIAL: NCT02792842
Title: Phase 2 Clinical Study of ART-123 for the Prevention of Cancer Treatment Related Symptoms in Patients With Postoperative Stage II / III Colon Cancer: a Multicenter Randomized Placebo-controlled Double-blind Study to Investigate the Efficacy and Safety of ART-123
Brief Title: Exploratory Study of ART-123 for the Prevention of Cancer Treatment Related Symptoms in Patients With Postoperative Stage II / III Colon Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ART-123-201
Record Dates: First submitted 2016-05-28; First posted 2016-06-08 (Estimated); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Stage II/III Colon Cancer
MeSH Terms: interventions — ART123

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- ART-123 (3-day ART) (Experimental)
  Interventions: Drug: ART-123 (3-day ART)
- ART-123 (1-day ART) (Experimental)
  Interventions: Drug: ART-123 (1-day ART)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ART-123 (3-day ART) — ART-123 380 U/kg infusion once daily on days 1-3 in each cycle
  Arms: ART-123 (3-day ART)
Drug: ART-123 (1-day ART) — ART-123 380 U/kg infusion once on day 1 and placebo infusion once daily on days 2-3 in each cycle
  Arms: ART-123 (1-day ART)
Drug: Placebo — Placebo infusion once daily on days 1-3 in each cycle
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ART-123 for the prevention of cancer treatment related symptoms in patients with postoperative stage II / III colon cancer.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosed with stage II / III colon cancer
* Deemed to have undergone curative A (Cur A) surgery
* Planning to undergo postoperative adjuvant chemotherapy

Main Exclusion Criteria:

* Have a history of hypersensitivity to any of the ingredients in thrombomodulin alfa (recombinant)
* Have any treatment history of systemic chemotherapy (including any drug in the clinical trial stage) or radiotherapy
* With active double cancer

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-07; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asahi Kasei Pharma Corporation, Study Chair — Asahi Kasei Pharma Corporation
Locations (2):
- Japan (2):
  - Kobe, Hyōgo
  - Nerima City, Tokyo

REFERENCES:
- [Derived] Kotaka M, Saito Y, Kato T, Satake H, Makiyama A, Tsuji Y, Shinozaki K, Fujiwara T, Mizushima T, Harihara Y, Nagata N, Kurihara N, Ando M, Kusakawa G, Sakai T, Uchida Y, Takamoto M, Kimoto S, Hyodo I. A placebo-controlled, double-blind, randomized study of recombinant thrombomodulin (ART-123) to prevent oxaliplatin-induced peripheral neuropathy. Cancer Chemother Pharmacol. 2020 Nov;86(5):607-618. doi: 10.1007/s00280-020-04135-8. Epub 2020 Sep 23. PMID 32965539

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ART-123 (3-day ART) | ART-123 (1-day ART) | Placebo
Started | 24 | 27 | 28
Completed | 20 | 23 | 21
Not Completed | 4 | 4 | 7
Not completed — Adverse Event | 4 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Schedule delay | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomly assigned participants who received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | ART-123 (3-day ART) | ART-123 (1-day ART) | Placebo | Total
Number analyzed (Participants) | 24 | 27 | 28 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 10 | 30
  >=65 years | 13 | 18 | 18 | 49
Age, Continuous [Median (Full Range); unit: years] | 66.0 [32 to 79] | 68.0 [38 to 78] | 68.0 [45 to 79] | 67.0 [32 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 12 | 40
  Male | 11 | 12 | 16 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 24 | 27 | 28 | 79

OUTCOME MEASURES:

1. Primary Outcome: The Cumulative Rates of Participants With NCI-CTCAE Grade 2 or Higher Peripheral Sensory Neuropathy: Up to End of Study Treatment
Description: NCI-CTCAE was used for investigator-reported outcomes of peripheral sensory neuropathy; it was assessed every day from day 1 to day 3 of each cycle and on days 15 (the day after 14 days have elapsed from the date of administration) of Cycle 12 and 43 (the day after 42 days have elapsed from the date of administration of Cycle 12) of cycle 12 as follow-up assessment. Once grade 2 or higher neuropathy was observed in a certain participant, that participant was categorized as grade 2 or higher even if the grade returned to 1 or lower in subsequent cycles. Participants who discontinued the study or whose evaluation data were missing without reaching grade 2 or higher neuropathy were analyzed as no grade 2 or higher neuropathy. No primary endpoint was specified due to the exploratory nature of the study.
Time Frame: 42 days after the start of cycle 12 (each cycle is 2 weeks).
Population: The preventive effect of ART-123 on neuropathy was analyzed in all randomly assigned participants who received at least one dose of study drug and oxaliplatin and had a FACT/GOG-Ntx-12 or NCI-CTCAE evaluation at least once after oxaliplatin administration.
Measure: Count of Participants; unit: Participants
Arm/Group | ART-123 (3-day ART) | ART-123 (1-day ART) | Placebo
Number analyzed (Participants) | 24 | 27 | 28
Participants | 11 | 11 | 18

2. Primary Outcome: Least-squares (LS) Means of Functional Assessment of Cancer Therapy/Gynecological Oncology Group-Neurotoxicity-12 (FACT/GOG-Ntx-12) Version 4.0 Score at Cycle 12
Description: Participant-reported outcomes were evaluated using the FACT/GOG-Ntx-12 version 4.0, which measured the severity and impact of symptoms of neuropathy over the past 7 days. Scores range from 0 to 48, with lower scores indicating more severe neurotoxicity. Participants completed paper questionnaires on days 1 and 8 of each cycle, on day 15 (the day after 14 days have elapsed from the date of administration) of cycle 12 and day 43 (the day after 42 days have elapsed from the date of administration) of cycle 12 as follow-up assessment. LS means were calculated from the mixed effect model for repeated measures (MMRM). Analysis included the fixed, categorical effects of study treatment, analysis visit, and study treatment-by-visit interaction. If multiple measurements occurred within the same visit, the measurement with the worst value was used. No primary endpoint was specified due to the exploratory nature of the study.
Time Frame: At baseline, at each cycle (up to cycle 12 with each cycle of 2 weeks), and follow-up assessment.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ART-123 (3-day ART) | ART-123 (1-day ART) | Placebo
Number analyzed (Participants) | 24 | 27 | 28
score on a scale | 32.3 [28.4 to 36.3] | 36.3 [32.4 to 40.1] | 28.9 [25.0 to 32.8]

3. Primary Outcome: The Discontinuation Rate of Oxaliplatin Due to Oxaliplatin-Induced Peripheral Neuropathy (OIPN)
Description: The number of people who discontinued oxaliplatin because of OIPN was counted and the percentage of the total was calculated. No primary endpoint was specified due to the exploratory nature of the study.
Time Frame: Cycle 12（each cycle is 2 weeks）
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ART-123 (3-day ART) | ART-123 (1-day ART) | Placebo
Number analyzed (Participants) | 24 | 27 | 28
Participants | 6 | 4 | 9

ADVERSE EVENTS:
Time Frame: From informed consent until the day 42 days have elapsed from the Cycle 12, with each cycle of 2 weeks, administration date
Arm/Group | ART-123 (3-day ART) | ART-123 (1-day ART) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 3/24 | 5/27 | 2/28
Other Adverse Events (participants affected / at risk) | 24/24 | 27/27 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ART-123 (3-day ART) (N=24) | ART-123 (1-day ART) (N=27) | Placebo (N=28)
Infective spondylitis (Infections and infestations) | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ART-123 (3-day ART) (N=24) | ART-123 (1-day ART) (N=27) | Placebo (N=28)
Nausea (Gastrointestinal disorders) | 9 | 12 | 9
Stomatitis (Gastrointestinal disorders) | 8 | 6 | 5
Constipation (Gastrointestinal disorders) | 4 | 7 | 6
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 5
Vomiting (Gastrointestinal disorders) | 2 | 2 | 4
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT02792842/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT02792842/SAP_001.pdf